CLINICAL TRIAL: NCT06299631
Title: Endoscopic Relapse Risk Factors After Ileocolic Resection on Crohn's Disease Patients in the Biologic Era
Brief Title: Endoscopic Relapse Risks Evaluation After Ileocolic Resection for Crohn's Disease
Acronym: RIC-1
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Carémeau University Hospital, Nîmes (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0187
Record Dates: First submitted 2023-11-29; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pathology sections blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohn's disease patients undergoing ICR: Crohn's disease patients undergoing ICR treated with TNF inhibitors
  Interventions: Procedure: Ileocolic resection

INTERVENTIONS:
Procedure: Ileocolic resection — Ileocolic resection by open or laparoscopic approach

SUMMARY:
Aim of the study:

To evaluate risk factors of endoscopic relapse after ileocolic resection in a cohort of Crohn's disease patients treated with anti-TNF agents.

Methods:

From 2014 to 2022, all consecutive patients who underwent ileocolic resection for Crohn's disease treated with anti-TNF agents in two referral tertiary center were prospectively collected.

Considering exclusion criteria, data from 114 patients were analyzed. The cohort was separated into 2 groups according to study period.

Short and long-term outcomes were compared between the two groups.

Primary outcome:

Endoscopic recurrence (defined as > i2 lesions according to Rutgeerts classification) 6 months after surgery

DETAILED DESCRIPTION:
Crohn's disease is a chronic inflammatory bowel disease whose preferential location is the ileo-colon, for which surgical management is necessary in 60% of patients.

The most common surgical procedure is ileo-caecal resection for symptomatic last ileal loop stenosis resistant to a well conducted medical treatment.

The conventional surgical technique aims to preserve the length of the digestive tract as much as possible. From a technical point of view, the resection passes as close as possible to the small intestine, leaving the vessels within the mesentery in place.

Despite the improvement of therapeutics (over the last decade, 80% of patients present an endoscopic recurrence at 1 year after surgery. Endoscopic recurrence is defined as the apparition of new typical mucosal lesions based on the Rutgeerts classification.

According to the last ECCO guidelines, biologic agents (TNF-inhibitors, ustekinumab and vedolizumab) are used as maintenance treatment in moderate-to-severe Crohn's disease patients:

* who achieved remission with anti-TNF agents -> maintenance treatment using the same treatment.
* who have achieved long-term remission with the combination of infliximab and immunosuppressants -> monotherapy with infliximab.
* who have achieved long-term remission with the combination of adalimumab and immunosuppressants -> monotherapy with adalimumab. The risk factors for postoperative recurrence are now well established and include smoking habit, penetrating or fistulizing phenotype (classified as B3 in the Montréal classification), perineal disease, history of previous bowel resection, extensive small bowel resection (>20 cm).

Recently, the role of the mesentery in Crohn's disease has been deeply investigated. There is a mesenteric nerve dysfunction with inhibition of anti-inflammatory activity, a major angiogenesis, a multiplication of lymphatic vessels with emboli at the origin of lymphatic drainage abnormalities, a mesenteric hypertrophy with multiple small adipocytes secreting adipokines.

These new elements have raised the question of a potential benefit of a combined resection of the mesentery during an ileocecal resection in the treatment of Crohn's disease.

CALVIN J Coffrey et al. carried out a study in 2008 comparing a prospective cohort with ileo-caecal resection including the mesentery (mesentery resection group) to a retrospective cohort with classical ileocecal resections (ICR group). The results were very promising in terms of recurrence requiring surgical management with a re-operation rate at 5 years of 40% in the classical ICR group vs 2.9% in the mesenteric resection group. And shows that significant mesenteric disease is an independent risk factor for recurrence with a HR=4.7 (p<0.007).

Thus, it is necessary to analyse within local patient base: the percentage of endoscopic recurrence at 6 months after surgery in patients treated with anti TNFa as well as the risk factors at the origin of the increase of these recurrences, more particularly the anatomopathological factors which could call into question the surgical practices within the long term a major interest in resection of the mesentery.

Therefore, the investigator carried out a retrospective study in two referral tertiary center, Montpellier University Hospital and Nîmes University Hospital. The investigator prospectively collected data from 2014 to 2022 from Crohn's disease patients treated with TNF inhibitors who have undergone ileocolic resection, to determine the percentage of endoscopic recurrence at 6 months and its risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven Crohn's disease
* On anti-TNF alpha: infliximab, adalimumab (ECCO 2014 recommendation)
* > 18 years old patients
* All patients who have undergone ileocolic resection and whose disease site is accessible to endoscopic follow-up (first or repeat procedure)

Exclusion Criteria:

* Minor patients under 18 years of age
* Endoscopic follow-up not possible
* Pregnant women
* Medical treatment other than anti-TNF alpha

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with Crohn's disease treated with TNF inhibitors who underwent ileocolic resection between 2014 and 2023 in the Digestive Surgery (A), Oncology and Minimally Invasive Department (Pr FABRE) of the Montpellier University Hospital and the Digestive Surgery and Cancer Department (Pr PRUDHOMME) of the Nimes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Endoscopic recurrence rate | 6 months after surgery
  Defined as the presenc of new mucosal lesions classified >i2 according to Rutgeerts classification.

SECONDARY OUTCOMES:
Resection margins | 90 days after surgery
  Pathological examination of resection margins
Length of resected specimen | 90 days after surgery
  Pathological examination and measure of the lenght of ileon and colon resection
Duration of surgery | 90 days after surgery
  Operative time
Intra-operative blood loss | 90 days after surgery
  Intra-operative blood losss
Postoperative morbidity rate | 90 days after surgery
  Postoperative morbidity according to Clavien Dindo
Mortality rate | 90 days after surgery
  Death occuring within 90 days after surgery
Myenteric plexitis | 90 days after surgery
  Myenteric plexitis defined as the presence of > 3 inflammatory cells in myenteric plexuses of the proximal resection margin
Number of inflammatory cells in myenteric plexuses | 90 days after surgery
  Number of inflammatory cells in myenteric plexuses of inflammatory cells in myenteric plexuses

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BARDOL, MD, MSc, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No